CLINICAL TRIAL: NCT06188247
Title: Pilot for a National Virtual Trial Testing Remote Sleep Apnea Evaluation in Patients with Atrial Fibrillation - (Mini VIR-SAAF)
Brief Title: Pilot-trial Testing Remote Sleep Apnea Evaluation in Patients with Atrial Fibrillation
Acronym: Mini VIR-SAAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Herlev and Gentofte Hospital (Other)
Responsible Party: Principal Investigator, Morten Lamberts, Associate Professor, Herlev and Gentofte Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2305474
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-01

CONDITIONS: Atrial Fibrillation; Sleep Apnea
MeSH Terms: conditions — Atrial Fibrillation; Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: NightOwl home-monitoring — The NightOwl™ system consists of a small sensor device which is placed on the fingertip and a smartphone app that is connected to an encrypted cloud-based analytics platform within the European Union, the NightOwl™ software. The sensor is self-applied by attaching the sensor to the fingertip by means of an adhesive patch. The NightOwl™ sensor acquires accelerometer data and reflectance-based photoplethysmography (PPG) from which it derives actigraphy (sleep/wake behavior), SpO2, peripheral artery tone (PAT) and pulse rate, among other features. A PAT analysis derives changes in caliber of arteries elicited by alterations in the contractile activity of vascular smooth muscle and are referred to as changes in arterial tone. The end state of the apnea-hypopnea events are associated with sympathetic activation.

SUMMARY:
This is an investigator-initiated virtual (or decentralized) trial that includes a postal parcel (mail-in) containing sensors for SA diagnosis (NightOwl™) and physical activity (SENS Motion), in addition to smart-phone based heart rhythm (FibriCheck) monitoring in participants with paroxysmal or persistent AF. A case-coordinator (the investigators) will manage all participant contacts virtually during the study from inclusion to follow-up.

DETAILED DESCRIPTION:
Objectives The main aim of the pilot trial is in a completely decentralized/virtual setting to evaluate whether SA home-evaluation, physical tracking by a home-monitoring device and heart rhythm monitoring by a smart-phone application in patients with AF are feasible.

Inclusion:

Confirmation of study eligibility will be performed entering key variables (including telephone number) into a secure web based program (RedCap) at the Cardiovascular Research Center at Herlev-Gentofte Hospital.

After inclusion, participants will receive a mail-in package containing the NightOwl™ device and the SENS Motion device. Online questionnaires for survey 1 will be pushed to participants via RedCap, which includes basic participant information (including mail, address, height, weight, (BMI), self-measured neck circumference and employment status) and the questionnaires Atrial Fibrillation Effect on QualiTy-of-life (AFEQT), AF severity scale (AFSS), Pittsburgh Sleep Quality Index (PSQI) and The eHealth Literacy Questionnaire (eHLQ).

Furthermore a clinical evaluation form will be filled out online in RedCap by the case coordinator based on electronic charts or from the video meeting which includes:

CPR number, sex, birthdate, questions related to AF: modified European Heart Rhythm Association (mEHRA) symptom classification (0-4), concomitant CVD medication (antithrombotic medication, rate-lowering drugs, anti-arrhythmic drugs, date of first AF detected, type of AF (paroxysmal or persistent AF), and other relevant medical conditions.

Postal Parcel 1:

After completing survey 1, a postal parcel (postal parcel 1) including the NightOwl device and the SENS Motion will be sent to the participant's address. The postal parcel 1 will also include detailed written information and instructions for the devices and applications together with a user-friendly written overview of the study design. As soon as the participants receive the postal parcel 1, the participant will begin their home monitoring with the 4 nights of NightOwl monitoring, the 7 days of activity tracker (round 1) with SENS Motion, and the heart rhythm monitoring with the FibriCheck application.

Return of equipment 1:

After completing the 4 nights of NightOwl monitoring and the 7 days of activity tracker round 1 with SENS Motion, the participants will ship the used SENS Motion and NightOwl device back to the case-coordinator. This will be done via a prepaid shipping label.

SA evaluation in cooperation with the Danish Center for Sleep Medicine, Glostrup:

Participants diagnosed with having a NightOwl evaluation showing moderate to severe SA (i.e. AHI>15) will be scheduled for a multidisciplinary meeting including case coordinator, SA specialist and cardiologist at site. At this meeting, the participant will be informed that the evaluation shows that significant SA is likely. Based on all information including patient symptoms, patient preferences and assessment by the multidisciplinary team, the following strategies is planned 1) fast-track initiation of remote CPAP treatment initiation 2) additional conventional SA work-up or CPAP treatment initiation at Glostrup Hospital, Copenhagen, 3) advice (e.g. sleep position trainer), or 4) no further investigation/treatment.

The strategy is based on clinical judgment. In case the assessment results in 1) or 2) the patient will be informed that a final diagnosis will be made by Dansk Center for Søvnsygdomme including the department will be responsible for any potential subsequent treatment.

Conventional SA work-up or CPAP treatment initiation In a subset of participants clinically selected for either a need for further clinically conventional SA workup or CPAP treatment, a referral to Danish Center for Sleep Medicine, Glostrup will be made.

The decision to either initiate treatment remotely or conventional is based on clinical judgment.

Postal Parcel 2:

At week 10, a postal parcel (postal parcel 2) with the SENS Motion will be sent to the participants' address for activity tracking (round 2). As soon as the participants receive the postal parcel 2, the participant will begin their 7 days of activity tracker round 2 with SENS Motion.

Return of equipment 2:

After completing the 7 days of activity tracker round 2 with SENS Motion, the participants will ship their used device back to the case-coordinator. This will be done via a prepaid shipping label.

Follow up:

After completing the 7 days of activity tracker round 2, questionnaires will once again be pushed digitally to participants including AFEQT, AFSS and PSQI. The questionnaires will be pushed again to participants a month after survey 2.

At week 12 the participant will be scheduled for a video meeting where the participant's own study results will be presented.

Evaluation: Qualitative interviews:

Finally, a subset of participants will be invited to focus-group interviews. One whole day workshop will be planned for evaluating major project elements (remote informed consent, eHealth literacy, digital device instructions, communication, multidisciplinary meeting and CPAP treatment, compliance). The evaluations will be used for identifying barriers for virtual trial inclusion, the use of devices and online completion of questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age>18 years
* Established paroxysmal or persistent AF diagnosis
* Owning a compatible smartphone (or accepting a smart phone provided by the investigators)
* Understanding of potential SA treatment possibilities including CPAP treatment

Exclusion Criteria:

* Previous investigation for sleep-disturbed breathing
* Advanced heart failure (left ventricular dysfunction and NYHA III/IV)
* Occupational driver licenses
* Pregnancy
* Doxazosin or Terazosin (alpha-adrenergic antagonists)
* Peripheral arterial disease with daily intermittent claudication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Drop-outs | 3 months
  The primary outcome of this pilot trial is the percentage of drop-outs (defined as not completing the 12 week study period) in participants given informed consent and having received the mail-in package.

CONTACTS AND LOCATIONS:
Locations (1):
- Herlev and Gentofte Hospital, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hashiba M, Al-Alak A, Nielsen SK, Kayser L, Nouhravesh N, Elmegaard M, El-Chouli M, Risom S, Frandsen RAV, Jennum P, Lamberts M. Feasibility of a decentralised trial of sleep apnoea screening in patients with atrial fibrillation. Dan Med J. 2025 Oct 2;72(11):A12240892. doi: 10.61409/A12240892. PMID 41133329